CLINICAL TRIAL: NCT02322762
Title: DISCOVERing Treatment Reality of Type 2 Diabetes in Real World Settings
Acronym: DISCOVER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00002
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Anti-diabetic management patterns
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One single cohort.: One single cohort of patients with type 2 diabetes mellitus initiating their second line anti-diabetic therapy after first line anti-diabetic therapy.

SUMMARY:
DISCOVER is a Non Interventional Study study to describe the disease management patterns and clinical evolution over three years in type 2 diabetes mellitus patients initiating a second line anti-diabetic treatment.

DETAILED DESCRIPTION:
DISCOVER is a NIS study to describe the disease management patterns and clinical evolution over three years in type 2 diabetes mellitus patients initiating a second line anti-diabetic treatment. This study is a multi-country, multicenter, observational, prospective, longitudinal cohort study. The patients will be recruitted from countries in Latin America, Europe and Asia pac. It is estimated that approximately 13350 patients will be enrolled in total with each patient followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of subject informed consent
2. Female or male aged 18 years and over
3. Diagnosed with type 2 diabetes mellitus
4. Initiating a second line anti-diabetic therapy, either as add-on, or switching from one monotherapy to another.

Exclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus
2. Patient is pregnant
3. Patients initiating a dual therapy after having previously received two different lines of monotherapy before (e.g.: Metformin → SU (Sulphonylureas) → SU+Add-on)
4. Current treatment with chemotherapy, oral or iv steroids
5. Patient is on dialysis or has had a renal transplant
6. The patient is taking insulin as first line treatment
7. The patient is taking dual therapy or a fixed dose combination treatment as first line treatment.
8. The patient is taking herbal remedies / natural medicines as first line treatment
9. Participation in an interventional trial
10. Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient for 3 years (e.g. lifethreatening co-morbidities, tourist, non-native speaker or does not understand the local language where interpreter services are not reliably available, psychiatric disturbances, dementia, alcohol or drug abuse).
11. Not willing to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus initiating their second line anti-diabetic therapy after first line anti-diabetic therapy. Participating investigators will belong to primary, secondary or tertiary care clinics or hospitals in proportions trying to resemble the reality of management of this type of patients in each country.
Sampling Method: Non-Probability Sample
Enrollment: 15992 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Anti-diabetic treatments prescribed by physicians in a real-world setting. | Up to 3 Years
  The drugs (or their combinations) prescribed by physicians to patients initiating a 2nd line anti-diabetic treatment in a real-world setting will be described at inclusion and during 3 years follow-up.

SECONDARY OUTCOMES:
Disease control in terms of achieving HbA1c target goals and reducing body weight and blood pressure. | Up to 3 years
Changes in anti-diabetic treatments | Up to 3 years
Disease progression (incidence of microvascular and macrovascular complications). | Up to 3 years
Incidence of hypoglycemic events. | Up to 3 years
Quality of Life, using Patient Reported Outcomes questionnaires. | Up to 3 years
Use of Healthcare resources. | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Medina, PhD, Study Director — AstraZeneca; Linong Ji, MD, Principal Investigator — Peking University People's Hospital, China; Bong Soo Cha, Dr., Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (303):
- Algeria (6):
  - Research Site, Algiers
  - Research Site, Batna City
  - Research Site, Blida
  - Research Site, Constantine
  - Research Site, Oran
  - Research Site, Sétif
- Argentina (9):
  - Research Site, Buenos Aires
  - Research Site, Chacabuco
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Paraná
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Australia (14):
  - Research Site, Blacktown
  - Research Site, Burwood
  - Research Site, Castle Hill
  - Research Site, Coorparoo
  - Research Site, Corio
  - Research Site, Cowra
  - Research Site, Edmonton
  - Research Site, Forbes
  - Research Site, Garran
  - Research Site, Ipswich
  - Research Site, Melbourne
  - Research Site, Sherwood
  - Research Site, Smithfield
  - Research Site, South Lake
- Austria (8):
  - Research Site, Feldbach
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Sankt Veit im Pongau
  - Research Site, Stankt Stefan Ob Stainz
  - Research Site, Vienna
- Research Site, Bahrain, Bahrain
- Brazil (13):
  - Research Site, Belo Horizonte
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Juiz de Fora
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, São José do Rio Preto
  - Research Site, São José dos Campos
  - Research Site, São Paulo
- China (22):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chenzhou
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hefei
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Nanjing
  - Research Site, Panjin
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shijiazhuang
  - Research Site, Shiyan
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Wuxi
- Colombia (5):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Manizales
  - Research Site, Medellín
- Costa Rica (3):
  - Research Site, Cartago
  - Research Site, Heredia
  - Research Site, San José
- Czechia (14):
  - Research Site, Benátky nad Jizerou
  - Research Site, Beroun
  - Research Site, Broumov
  - Research Site, Dolní Břežany
  - Research Site, Karlovy Vary
  - Research Site, Krnov
  - Research Site, Litoměřice
  - Research Site, Náchod
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Uherské Hradiště
  - Research Site, Újezd u Brna
- Egypt (8):
  - Research Site, Al Mansurah
  - Research Site, Alexandria
  - Research Site, Asyut
  - Research Site, Cairo
  - Research Site, Giza
  - Research Site, Heliopolis
  - Research Site, Minya
  - Research Site, Tanta
- India (19):
  - Research Site, Bangalore
  - Research Site, Chandigarh
  - Research Site, Chennai
  - Research Site, Coimbatore
  - Research Site, Delhi
  - Research Site, Ghaziabad
  - Research Site, Gūrgaon
  - Research Site, Hyderabad
  - Research Site, Indore
  - Research Site, Jaipur
  - Research Site, Kanpur
  - Research Site, Karnāl
  - Research Site, Kolkata
  - Research Site, Mangalore
  - Research Site, Mumbai
  - Research Site, Nagpur
  - Research Site, Noida
  - Research Site, Pune
  - Research Site, Trivandrum
- Indonesia (9):
  - Research Site, Balikpapan
  - Research Site, Banda Aceh
  - Research Site, Batu
  - Research Site, Bekasi Timur
  - Research Site, Denpasar
  - Research Site, Jakarta
  - Research Site, Malang
  - Research Site, Manado
  - Research Site, Padang
- Italy (11):
  - Research Site, Foggia
  - Research Site, Garbagnate Milanese
  - Research Site, Livorno
  - Research Site, Mariano Comense
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Potenza
  - Research Site, Rimini
  - Research Site, Roma
  - Research Site, Sesto San Giovanni
- Jordan (3):
  - Research Site, Amman
  - Research Site, Az Zarqaa
  - Research Site, Irbid
- Research Site, Kuwait City, Kuwait
- Lebanon (8):
  - Research Site, Beirut
  - Research Site, Byblos
  - Research Site, Chtoura
  - Research Site, Hamra
  - Research Site, Mazraat Yachouaa
  - Research Site, Saida
  - Research Site, Tripoli
  - Research Site, Tyre
- Malaysia (11):
  - Research Site, Alor Star
  - Research Site, Ayer Itam
  - Research Site, Ipoh
  - Research Site, Johor Bahru
  - Research Site, Kelantan
  - Research Site, Kuala Krai
  - Research Site, Masjid Tanah
  - Research Site, Miri
  - Research Site, Perak
  - Research Site, Sandakan
  - Research Site, Seremban
- Mexico (9):
  - Research Site, Acapulco de Juárez
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, San Juan del Río
  - Research Site, Tamaulipas
  - Research Site, Zapopan
- Netherlands (32):
  - Research Site, Almelo
  - Research Site, Alpen Aan Den Rijn
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, De Bilt
  - Research Site, Doetinchem
  - Research Site, Dordrecht
  - Research Site, Dorst
  - Research Site, Elst
  - Research Site, Enschede
  - Research Site, Etten-Leur
  - Research Site, Garderen
  - Research Site, Geleen
  - Research Site, Gouda
  - Research Site, Hoogezand
  - Research Site, Katwijk
  - Research Site, Kerkrade
  - Research Site, Kloosterhaar
  - Research Site, Landgraaf
  - Research Site, Luttenberg
  - Research Site, Nijverdal
  - Research Site, Oisterwijk
  - Research Site, Roermond
  - Research Site, Soerendonk
  - Research Site, Steenbergen
  - Research Site, The Hague
  - Research Site, Utrecht
  - Research Site, Vaassen
  - Research Site, Voerendaal
  - Research Site, Wamel
  - Research Site, Zoetermeer
  - Research Site, Zundert
- Research Site, Muscat, Oman
- Panama (2):
  - Research Site, Calle
  - Research Site, Coclé
- Poland (11):
  - Research Site, Chorzów
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Parczew
  - Research Site, Rzeszów
  - Research Site, Zabrze
  - Research Site, Zgierz
- Russia (11):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Sestroretsk
  - Research Site, Stavropol
  - Research Site, Yaroslavl
- Saudi Arabia (5):
  - Research Site, Abhā
  - Research Site, Al Jouf
  - Research Site, Jeddah
  - Research Site, Khamis Mushait
  - Research Site, Riyadh
- South Africa (11):
  - Research Site, Alberton
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Johannesburg
  - Research Site, Lenasia
  - Research Site, Merebank
  - Research Site, Midstream
  - Research Site, Moloto South
  - Research Site, Port Elizabeth
  - Research Site, Pretoria
- South Korea (10):
  - Research Site, Bucheon-si
  - Research Site, Cheonan-si
  - Research Site, Chuncheon
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Gwangmyeong
  - Research Site, Iksan
  - Research Site, Jeju Special Self-Governing Province
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (11):
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Elche
  - Research Site, Espinardo
  - Research Site, Madrid
  - Research Site, Móstoles
  - Research Site, Salamanca
  - Research Site, Sanlúcar de Barrameda
  - Research Site, Segovia
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Tunisia (11):
  - Research Site, Gabès
  - Research Site, Kairaouane
  - Research Site, Mahdia
  - Research Site, Montfleury
  - Research Site, Mutuelleville
  - Research Site, Nabeul
  - Research Site, Sfax
  - Research Site, Sousse
  - Research Site, Sukrah
  - Research Site, Tunis
  - Research Site, Tunis Belvedere
- Turkey (Türkiye) (16):
  - Research Site, Adana
  - Research Site, Afyonkarahisar
  - Research Site, Antalya
  - Research Site, Çanakkale
  - Research Site, Çorum
  - Research Site, Denizli
  - Research Site, Diyarbakır
  - Research Site, Düzce
  - Research Site, Elâzığ
  - Research Site, Gaziantep
  - Research Site, Hatay
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Karaman
  - Research Site, Kayseri
  - Research Site, Samsun
- United Arab Emirates (2):
  - Research Site, Abu Dhabi
  - Research Site, Dubai

REFERENCES:
- [Derived] Al Rubeaan K, Banah F, Alruwaily FG, Sheshah E, Alnaqeb D, AlQahtani AM, Ewais D, Al Juhani N, Hassan AH, Youssef AM. Metabolic control and incidence of hypoglycaemia, hospitalisation and complications among Saudi patients with type 2 diabetes initiating second-line therapy: an analysis of the Saudi Arabia data from the DISCOVER Observational Study programme. BMJ Open. 2023 Aug 30;13(8):e063586. doi: 10.1136/bmjopen-2022-063586. PMID 37648382
- [Derived] Al-Rubeaan K, Banah F, Alruwaily FG, Sheshah E, Alnaqeb D, AlQahtani AM, Ewais D, Al Juhani N, Hassan AH, Youssef AM. Longitudinal assessment of the quality of life and patterns of antidiabetic medication use in patients with type 2 diabetes, Saudi Arabia perspective, DISCOVER study. Curr Med Res Opin. 2023 Jan;39(1):27-35. doi: 10.1080/03007995.2022.2144052. Epub 2022 Nov 28. PMID 36342972
- [Derived] Mita T, Katakami N, Takahara M, Kawashima M, Wada F, Akiyama H, Morita N, Kidani Y, Yajima T, Shimomura I, Watada H. Changes in Treatment Satisfaction Over 3 Years in Patients With Type 2 Diabetes After Initiating Second-line Treatment. J Clin Endocrinol Metab. 2022 Aug 18;107(9):2424-2432. doi: 10.1210/clinem/dgac420. PMID 35857060
- [Derived] Hejjaji V, Gorgojo-Martinez JJ, Tang F, Garnelo JB, Cooper A, Medina J, Mutiozabal MS, Khunti K, Nicolucci A, Shestakova MV, Ji L, Gomes MB, Watada H, Vora J, Malik AO, Kosiborod M, Arnold SV. Factors associated with weight loss in people with overweight or obesity living with type 2 diabetes mellitus: Insights from the global DISCOVER study. Diabetes Obes Metab. 2022 Sep;24(9):1734-1740. doi: 10.1111/dom.14745. Epub 2022 May 25. PMID 35546275
- [Derived] Khunti K, Gomes MB, Kosiborod M, Nicolucci A, Pocock S, Rathmann W, Shestakova MV, Shimomura I, Watada H, Chen H, Cid-Ruzafa J, Fenici P, Hammar N, Tang F, Ji L; DISCOVER Scientific Committee and all DISCOVER investigators. Metformin discontinuation in patients beginning second-line glucose-lowering therapy: results from the global observational DISCOVER study programme. BMJ Open. 2020 Aug 30;10(8):e034613. doi: 10.1136/bmjopen-2019-034613. PMID 32868349
- [Derived] Wang JS, Chen H, Tang F, Sheu WH. Associations of fear of hypoglycemia with second-line use of insulin secretagogues or insulin and subsequent glycemic control in patients with type 2 diabetes: An analysis using data from the DISCOVER study. Int J Clin Pract. 2020 Jun;74(6):e13485. doi: 10.1111/ijcp.13485. Epub 2020 Feb 11. PMID 32003099
- [Derived] Khunti K, Chen H, Cid-Ruzafa J, Fenici P, Gomes MB, Hammar N, Ji L, Kosiborod M, Pocock S, Shestakova MV, Shimomura I, Tang F, Watada H, Nicolucci A; DISCOVER investigators. Glycaemic control in patients with type 2 diabetes initiating second-line therapy: Results from the global DISCOVER study programme. Diabetes Obes Metab. 2020 Jan;22(1):66-78. doi: 10.1111/dom.13866. Epub 2019 Oct 1. PMID 31468637
- [Derived] Nicolucci A, Charbonnel B, Gomes MB, Khunti K, Kosiborod M, Shestakova MV, Shimomura I, Watada H, Chen H, Cid-Ruzafa J, Fenici P, Hammar N, Surmont F, Tang F, Pocock S. Treatment patterns and associated factors in 14 668 people with type 2 diabetes initiating a second-line therapy: Results from the global DISCOVER study programme. Diabetes Obes Metab. 2019 Nov;21(11):2474-2485. doi: 10.1111/dom.13830. Epub 2019 Aug 5. PMID 31297947
- [Derived] Khunti K, Ji L, Medina J, Surmont F, Kosiborod M. Type 2 diabetes treatment and outcomes worldwide: A short review of the DISCOVER study programme. Diabetes Obes Metab. 2019 Nov;21(11):2349-2353. doi: 10.1111/dom.13817. Epub 2019 Jul 14. PMID 31215715
- [Derived] Kosiborod M, Gomes MB, Nicolucci A, Pocock S, Rathmann W, Shestakova MV, Watada H, Shimomura I, Chen H, Cid-Ruzafa J, Fenici P, Hammar N, Surmont F, Tang F, Khunti K; DISCOVER investigators. Vascular complications in patients with type 2 diabetes: prevalence and associated factors in 38 countries (the DISCOVER study program). Cardiovasc Diabetol. 2018 Nov 28;17(1):150. doi: 10.1186/s12933-018-0787-8. PMID 30486889
- See also: redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690R00002&attachmentIdentifier=d1e8378e-8782-4201-9b0e-72debb1b124c&fileName=DISCOVER_study_report_synopsis_redacted.pdf&versionIdentifier=